CLINICAL TRIAL: NCT02674256
Title: The Effect of Corticotrophin-releasing Hormone (CRH) on Esophageal Sensitivity in Healthy Volunteers: A Randomized, Single-blind, Placebo-controlled Study
Brief Title: The Effect of Corticotrophin-releasing Hormone (CRH) on Esophageal Sensitivity in Healthy Volunteers
Acronym: CRH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: S56177
Record Dates: First submitted 2014-03-25; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Sensitivity (Hyper); Gastrointestinal
Keywords: health; age between 18 to 60 years old; no history of gastrointestinal symptoms or complaints
MeSH Terms: conditions — Hypersensitivity | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRH injection (Active Comparator): Intervention: intravenous injection of CRH 100µg CRH powder for injection (CRH ferring®, Ferring, Aalst, Belgium) and 1 mL of NaCl 0.9% will be put together then the solution will be injected IV over the course of 1 minute
  Interventions: Drug: CRH
- placebo injection (Placebo Comparator): Intervention: intravenous saline injection
  1mL of saline will be injected intravenously over the course of 1 minute
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CRH — 100µg CRH powder for injection (CRH ferring®, Ferring, Aalst, Belgium) and 1 mL of NaCl 0.9% will be put together, then the solution will be injected intravenously over the course of 1 minute
  Other Names: CRH ferring®, Ferring, Aalst, Belgium
  Arms: CRH injection
Other: Placebo — 1 mL of NaCl 0.9% will be injected intravenously over the course of one minute
  Other Names: Saline solution
  Arms: placebo injection

SUMMARY:
Introduction and aim

Stress is well known to affect visceral sensitivity in Human. The investigators speculate that visceral hypersensitivity plays an important role in symptom perception in gastro-esophageal reflux disease (GERD). The role of acute stress mimicked by corticotrophin releasing hormone (CRH) administration on esophageal sensitivity has not been studied. The investigators hypothesize that stress mediated through CRH-release increases esophageal sensitivity. A first step in the investigation of this hypothesis is to study whether administration of CRH has an influence on esophageal sensitivity in healthy volunteers (HV). Therefore, the aim of this study is to investigate the effect of CRH-administration on esophageal sensitivity in a group of HV.

Methods

The study will be performed in cross-over on 15 HV with no prior history of digestive disease. Esophageal sensitivity will be tested by multimodal stimulation on two sessions (placebo and CRH-administration), with an interval at least of one week. The two sessions will be scheduled by randomization for every subject. After blinded administration of CRH 100µg or placebo IV, esophageal sensitivity will be assessed using a multimodal esophageal stimulation probe which allows thermal, mechanical, electrical and chemical stimulations of the esophagus. Esophageal sensitivity will be assessed using Visual Analogue Scale (VAS), the mood with specific questionnaires (Manikin Self assessment SAM, Profile of Mood Schedule (POMS, State Trait Anxiety Inventory (STAI)) and the cortisol with salivary samples.

Statistical analysis

Esophageal sensitivity for the different stimuli (heat, mechanical, electrical and chemical) will be compared between CRH and placebo conditions. To determine the stress-inducing capability of CRH-administration, the POMS questionnaire, STAI, Manikin self assessment and cortisol levels after the stress-protocol will be compared with the basal measurements.

Perspectives

If CRH-administration increases esophageal sensitivity, a stress model could be applied to investigate the influence of a real life stressor on esophageal sensitivity in healthy subjects. In a third part, a mast-cell stabilizing drug could be tested after administration of a stressor in order to investigate its role on esophageal sensitivity. In the future, this might be proposed to refractory GERD in a controlled randomized trial.

DETAILED DESCRIPTION:
1. INTRODUCTION Gastro-esophageal reflux disease (GERD) is the presence of symptoms (heartburn, regurgitation) or lesions that can be attributed to the reflux of gastric contents into the esophagus. In humans, pain is a multimodal experience composted of sensory, physiological and psychological aspects. In order to mimic the clinical situation, experimental models should be based on multimodal testing regimens in which different receptors and central nervous system mechanisms are activated. Typical and atypical symptoms may not only arise from acid reflux, but also from reflux with less acidic pH (pH 4-7). In GERD patients with persisting symptoms on proton pump inhibitor (PPI) therapy, ongoing weakly acidic reflux is well established as an important underlying factor. The basis for symptom generation during weakly acidic reflux remains to be determined, but acid sensitivity in the pH range 4-7, mechanical distension, sensitivity to other chemical factors and esophageal hypersensitivity to physiological levels of reflux have been proposed. The investigators speculate that visceral hypersensitivity plays an important role in symptom perception. This is suggested by the reflux parameters that are usual within the physiological number during PPI therapy. Also, the investigators previously demonstrated that refractory GERD patients have increased visceral hypersensitivity for thermal, chemical and mechanical esophageal stimulation compared to HV.

   Stress is well known to affect visceral sensitivity in humans. A majority of patients with GERD report stress as an important factor triggering symptom exacerbation. A real-life stressor could exacerbate heartburn in GERD patients by enhancing perceptual response to esophageal acid exposure. The interaction between psychological state and GI function is a complex and developing field. The brain-gut axis, mediating the effects of stress on the Gastrointestinal (GI) tract, has been considered a pivotal player in the pathogenesis of functional GI disorders like irritable bowel syndrome (IBS) and functional dyspepsia (FD). A possible mechanism of stress-induced visceral sensitivity could be the barrier dysfunction. A study performed in humans, showed that an acute psychological stressor induces hyperpermeability in a mast cell dependent fashion and exogenous peripheral CRH recapitulated its effects on barrier function. This increase in intestinal permeability is a phenomenon which appears as a prerequisite for visceral hypersensitivity. The acute role of CRH on esophageal sensitivity has not been studied.
2. OBJECTIVE Stress increases permeability via CRH-mediated mast cell activation. The investigators hypothesize that stress mediated through CRH-release increases esophageal sensitivity. Therefore, the aim of our study is to investigate the effect of CRH-administration on esophageal sensitivity in a group of HV.
3. GENERAL DESCRIPTION Studies will be performed in HV. All participants will receive and sign a copy of the informed consent before initiation of the study. Esophageal sensitivity will be tested by multimodal stimulation on two sessions (placebo and CRH-administration).
4. MATERIALS AND METHODS Studies will be performed using a multimodal esophageal stimulation probe which allows esophageal thermal, mechanical, electrical and chemical stimulations.

   During each stimulation, HV will record symptom perception using VAS. First perception (VAS=1), pain perception threshold (VAS=5) and pain tolerance threshold (VAS=7) will be recorded. All stimulations will be immediately terminated when the VAS 7 is reached. At the time of VAS 7, subjects will be asked to draw the referred pain area, to identify pain location.

   Thermal stimulation will be performed by re-circulating a saline solution, heated by a water bath, through the balloon mounted on the probe. Stimulation temperature will be steadily increased by increasing the flow rate from the water bath to the balloon. The volume in the balloon will be kept constant (5ml) to avoid mechanical stimulation. A temperature sensor in the balloon will continuously monitor the stimulation temperature, which is displayed online on a computer throughout the study.

   Mechanical stimulation will be performed by distension of the balloon. The flow of saline into the balloon, inducing the distension, is regulated by a computer controlled pump. The volume in the balloon is displayed on the computer screen throughout the stimulation. Mechanical stimulations will be performed with water of 37 degrees Celsius, to avoid thermal stimulation.

   Electrical stimulation will be performed by 2 electrodes mounted on the probe. Single burst pulses will be given with duration of 1ms at 200Hz. The amplitude of the pulses will increase with steps of 0.5mA. The maximum intensity is limited to 50 mA, as previous studies have shown atrial capturing with higher intensities. Electrocardiogram (ECG) monitoring will be performed as a safety measure during the electrical stimulations.

   Chemical stimulation will be performed by infusing an acidic solution (HCl 0.1N) in the distal esophagus, with a flow rate of 2ml/min. The stimulation will last for a maximum of 30 min.

   After an overnight fast subjects will come to the endoscopy unit of the Universitary Hospital of Leuven,Gasthuisberg, where the study will be performed. Two sessions will be scheduled for every subject: one placebo and one CRH session, with one week interval at least between each of them. Sessions will run in a single-blind way, as far as the placebo or drugs are concerned. The order of placebo and CRH-administration will be randomized by drawing cards from a box of cards determining the sequence.

   At the beginning of the session, the multimodal stimulation probe will be positioned through the mouth. After the probe is positioned in the esophagus, it will be fixed to the chin and the subject will remain in semi-recumbent position for the entire study. Before the actual stimulations start, there will be an adaptation period of 15 min, to get used to the feeling of the probe and to provide instructions for the correct use of the VAS meter. Fifteen minutes after the ingestion of the multimodal esophageal stimulation probe, 100µg CRH powder for injection (CRH ferring®, Ferring, Aalst, Belgium) and 1mL of NaCl 0.9% will be put together, then the solution will be injected intravenously over the course of 1 minute. With this dose, side-effects are limited to transient facial flushing that lasts from 5 to 45 min in 75% of patients. During placebo sessions, 1mL of NaCl 0.9% will be put in an identical syringe as the one used for CRH administration, and then injected intravenously (IV). In this way the HV will be blinded for the administration of CRH or placebo. Over time, each HV will receive placebo or CRH in the first session in a random sequence. In the second session, the subject will receive the other product that he/she didn't receive the first time.

   Salivary samples will be obtained at each session to determine salivary cortisol immediately before placebo or CRH-administration, at 30, 60, 90 and 120 min after administration. Salivary cortisol will be determined by ELISA. On every session, an assessment of general mood will be performed by the POMS and the STAI state questionnaires before and after the stimulation tests. The POMS consists of words describing different feelings and emotions at the present moment. The STAI state is validated, and widely used measuring transitory anxiety states.
5. DATA ANALYSIS The main objective is to show a difference for thermal stimulation with or without injection of CRH. The number of HV to be included is calculated with a medium comparison test. For a first species of risk α of 5% and a unilateral formulation, the investigators need to include 15 HV in total in order to highlight the expected differences and ensure a power of 80%.

   Temperature, volume, cross-section area of the balloon, pressure and electrical current will be measured at first perception, pain perception threshold and pain tolerance threshold and will be used to determine esophageal sensitivity. Esophageal sensitivity for the different stimuli (heat, mechanical, electrical and chemical) will be compared between CRH and placebo conditions.

   To determine the stress-inducing capability of CRH-administration, the POMS, STAI and cortisol levels after the stress-protocol will be compared with the basal measurements of the first study day.
6. PERSPECTIVES If CRH-administration increases esophageal sensitivity, a stress model could be applied to investigate the influence of a real life stressor on esophageal sensitivity in HV. In a third part, a mast-cell stabilizing drug could be tested after administration of a stressor in order to investigate its role on esophageal sensitivity. In the future, this might be proposed to refractory GERD in a controlled randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* age between 18 to 60 years

Exclusion Criteria:

* no history of gastrointestinal symptoms or complaints
* history of allergic reaction to CRH
* pregnancy or lactation
* concomitant administration of monoamine oxidase inhibitors (MAOI), verapamil or diltiazem or medication affecting esophageal motility
* significant co-morbidities (neuromuscular, psychiatric, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic)
* prior history of esophageal, ENT or gastric surgery or endoscopic anti-reflux procedure
* history of gastrointestinal disease and first degree relatives with Crohn's disease or celiac disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measurement of changes in esophageal sensitivity after IV CRH administration | 2 sessions per HV with at least one week interval, duration of each session: approximately 2 hours and 30 minutes. Temperature stimulation: 30 minutes
  Investigation of the effect of CRH-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the Temperature values (°C) of the stimulation tests between the placebo and CRH condition to see if CRH affects the sensitivity to increasing temperature.
Measurement of changes in esophageal sensitivity after IV CRH administration | 2 sessions per HV with at least one week interval, duration of each session: approximately 2 hours and 30 minutes. Mechanical stimulation: 30 minutes
  Investigation of the effect of CRH-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the balloon volumes (volume in ml) of the stimulation tests between the placebo and CRH condition to see if CRH affects the sensitivity to increasing balloon volume.
Measurement of changes in esophageal sensitivity after IV CRH administration | 2 sessions per HV with at least one week interval, duration of each session: approximately 2 hours and 30 minutes. Electrical stimulation: 30 minutes
  Investigation of the effect of CRH-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the tolerated intensity of the electrical pulses (mA) of the stimulation tests between the placebo and CRH condition to see if CRH affects the sensitivity to increasing electrical pulses.
Measurement of changes in esophageal sensitivity after IV CRH administration | 2 sessions per HV with at least one week interval, duration of each session: approximately 2 hours and 30 minutes. Chemical stimulation: 30 minutes
  Investigation of the effect of CRH-administration on esophageal sensitivity to multimodal stimulation in a group of healthy volunteers. This will be assessed by comparing the volume of infused acid (ml) of the stimulation tests between the placebo and CRH condition to see if CRH affects the sensitivity to acid infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Tack, MD, PhD, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No